CLINICAL TRIAL: NCT06211010
Title: The Urinary Cancer Detection by the Target Urine Volatile Organic Compounds Biosensor
Brief Title: The Target Urine VOCs Biosensor for Genitourinary Malignancy Detection
Status: Completed | Type: Observational
Sponsor: Suranaree University of Technology (Other)
Responsible Party: Principal Investigator, CHATCHAI, Associate Professor Dr. Chatchai Kreepala, M.D., Suranaree University of Technology
Other Study IDs: EC-64-109
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: The Phenomenon of the Decrease in the Electrical Resistance Within the Conducting Chambers, Making the Increase in a Conducting Property
Keywords: Volatile Organic Compounds (VOCs); Biosensor; Genitourinary Cancer
MeSH Terms: conditions — Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Fresh Urine sample 20 mL for a pateint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the semiconductor metal oxide sensors. — The method of analyzing the VOCs was through analyzing the evaporated VOCs from the urine in the container when they evaporated into the sealed chamber. The VOCs in the chamber were then analyzed at the same time by the five different gas semiconductor sensors which were located on the top of the chamber.
  Other Names: The detailed products and basic semiconductor circuits are available in the Figaro Product Information Manual (https://www.figarosensor.com/product/sensor/).

SUMMARY:
Volatile organic compounds (VOCs) have grown due to their crucial role in transitioning from invasive to noninvasive cancer diagnostic methods. This study aimed to assess the feasibility of the metal oxide biosensor platform using urine VOCs for detecting genitourinary cancers.

Five different commercially available semiconductor sensors were chosen to detect specific VOCs (methane, iso-butane, hydrogen, ethanol, hydrogen sulfide, ammonia, toluene, butane, propane, trimethylamine, and methyl-mercaptan). Changes in electrical resistance due to temperature variations from the voltage heater were examined to characterize VOC metabolism. Logistic regression and ROC analysis were employed to evaluate potential urine VOCs for genitourinary cancer determination.

DETAILED DESCRIPTION:
Nowadays, the development of semiconductor metal oxide sensors allows the detection of VOCs from breath and urine by relying on the change of voltage and electrical resistance. The studies use electric current to evaporate VOCs and focus on the changes of evaporation at different temperatures. The results from the previous studies have shown that the changes in the voltage and electrical current resistance dynamics in the semiconductor metal oxide sensors indicate specific patterns that are specific to different types of VOCs. Therefore, this could transit the odor-fingerprint in biogas expression platform to the electrical expression platform due to the possibility of specific-disease VOC identification and the cost-effectiveness of the electrical expression platform when compared to SPME and GC-MS.

This is a descriptive cohort study conducted among 64 subjects attending outpatient clinic at during August 2021 to July 2023. All the subjects were advised and voluntarily signed a consent form before participating in our study. The patients with the renal diseases and the normal subjects were prohibited to have strong odor food (such as tea, coffee, onion, garlic, shrimp paste, acacia, fermented fish, pakria, and celery, etc.) for at least 3 hours before the examination of urine VOCs and were prohibited alcohol intakes for more than 24 hours prior to the urine VOCs examination. The urine samples were collected for 20 mL in universal bottles and samples were classified as genitourinary (kidney/bladder/prostate) cancer or non-cancer or normal control after pathological examination of the biopsy specimens. The urine samples were kept at room temperature and taken to be analyzed with the semiconductor sensors within 30 minutes after the samples were collected.

We selected five different commercially available semiconductor metal oxide sensors to detect all the targeted VOCs, which are methane, iso-butane, hydrogen, ethanol, hydrogen sulfide, ammonia, toluene, butane, propane, trimethylamine, methyl-mercaptan (manufactured by Figaro company). These are the types of VOCs which had been studied and were shown to be related to the malignant according to the literature. The detailed products and basic semiconductor circuits are available in the Figaro Product Information Manual (https://www.figarosensor.com/product/sensor/).

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years

Exclusion Criteria:

* The patients with the renal diseases and the normal subjects were prohibited to have strong odor food

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pateints at Nephrology and Urology clinic of Suranaree University of Technology
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
the Target Urine Volatile Organic Compounds from urinary cancers | DEC 2021-SEP 2023
  urine VOCs for detecting genitourinary cancers

CONTACTS AND LOCATIONS:
Overall Officials: Chatchai Kreepala, M.D., Principal Investigator — School of Internal Medicine, Institute of Medicine, Suranaree University of Technology, Thailand
Locations (1):
- Institute of Medicine, Suranaree University of Technology, Nakhon Ratchasima, Thailand

IPD SHARING:
Plan to Share IPD: No
pateints' name and hospital numbers were not indebtifed.